CLINICAL TRIAL: NCT00167024
Title: Application of Genetic Polymorphisms of DNA Repair in The Prediction of Prostate Cancer Susceptibility and Its Clinical Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700307
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2005-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer, DNA repair gene, genetic polymorphism
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Primary: to investigate the effects of DNA repair gene polymorphisms on prostate cancer susceptibility, pathological grade, disease stage and clinical outcome Secondary: to understand the association between DNA repair gene polymorphism and prostate cancer and provided important information for screening, prevention and treatment of prostate cancer

DETAILED DESCRIPTION:
DNA repair plays a key role in carcinogenesis through the removal and repair of DNA damage induced by endogenous and environmental sources. The DNA repair system included four pathways: 1) Base Excision Repair (BER), 2) Nucleotide Excision Repair (NER), 3) Mismatch Repair (MMR) and 4) Double-Strand Break Repair, including homologous recombination pathway and nonhomologous end-joining repair pathway. Decreased and impaired DNA repair capacity has been reported in various cancers, however, its effect on prostate cancer still under investigated.

Common polymorphisms in DNA repair gene may alter protein function and individual's capacity to repair damaged DNA, hence, influence the cancer susceptibility. Polymorphic variants of DNA repair gene have been found to be associated with cancer susceptibility, but rare studies have investigated their effect on prostate cancer. Since variation in the function of these DNA repair genes also impact a cancer cell's viability or resistance to treatment, genetic variants in DNA repair might serve as a valuable biomarker in forcasting the result of cancer treatment. In fact, some reports have demonstrated the association between polymorphisms of DNA repair genes and results of treatment of various cancers.

For the present study proposal, we focused on several DNA repair genes: X-ray repair cross- complementing group 1 (XRCC1), human oxoguanine glycosylase I (hOGG1), xeroderma pigmentosum complementation group D (XPD), hMSH2, hMLH1 and X-ray repair cross-complementing group 3 (XRCC3), which might have relevance in prostate carcinogenesis based on their known functions. XRCC1 is involved in DNA repair in the base excision pathway, the hOGG1 gene encodes a DNA glycosylase /apurinic-apyrimidinic lyase that catalyzes the excision and removal the 8-OH-dG (8-hydroxy- 2-deoxyguanine) - which is a major form of oxidative DNA damage. The XPD gene codes for a DNA helicase involved in transcription and nucleotide excision repair. The hMSH2 and hMLH1 are genes involved with mismatch repair. The XRCC3 gene encoded a protein in the double-strand break homologous recombinational repair pathways.

In this proposed study, we will also use PCR-based methods to investigate the effects of DNA repair gene polymorphisms on prostate cancer susceptibility, pathological grade, disease stage and clinical outcome. With these efforts, we will further understand the association between DNA repair gene polymorphism and prostate cancer and provided important information for screening, prevention and treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer approved by pathology

Exclusion Criteria:

* combined with other malignancy
* accepting blood transfusion within 6 months

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Yuan Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan